CLINICAL TRIAL: NCT03311308
Title: Profiling and Reversing Metabolic Insufficiency in the Tumor Microenvironment in Advanced Melanoma: A Trial of Pembrolizumab and Metformin Versus Pembrolizumab Alone in Advanced Melanoma
Brief Title: A Trial of Pembrolizumab and Metformin Versus Pembrolizumab Alone in Advanced Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yana Najjar (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Yana Najjar, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 16-196
Record Dates: First submitted 2017-09-18; First posted 2017-10-17 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Advanced Melanoma
Keywords: Melanoma; Unresectable; Stage III; Stage IV
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab (Active Comparator): Pembrolizumab (Keytruda), 200 mg, by IV, every three weeks, for up to 2 years; after the first three doses, dosing can be changed to 400mg IV every 6 weeks, at the treating physician's discretion.
  Interventions: Drug: Pembrolizumab Injection [Keytruda]
- Pembrolizumab and Metformin Combination (Experimental): Pembrolizumab (Keytruda), 200mg, by IV, every three weeks, for up to 2 years will be taken in combination with Metformin, 500mg, twice a day, for nine weeks; after the first three doses, pembrolizumab dosing can be changed to 400mg IV every 6 weeks, at the treating physician's discretion.
  Interventions: Drug: Pembrolizumab Injection [Keytruda]; Drug: Metformin

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — 200mg, IV, every three weeks, up to two years; After the first three doses, dosing can be changed to 400mg IV every 6 weeks, at the treating physician's discretion.
  Other Names: Keytruda
Drug: Metformin — 500 mg, by mouth, twice a day for nine weeks.
  Arms: Pembrolizumab and Metformin Combination

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the combination of Pembrolizumab (KEYTRUDA®) and the investigational drug, Metformin.

DETAILED DESCRIPTION:
Patients are being asked to take part in this clinical research study because they have advanced, un-resectable stage III or IV Melanoma. If they participate they will be randomized to receive Pembrolizumab (KEYTRUDA®) or the combination of Pembrolizumab (KEYTRUDA®) plus Metformin.

This research study will evaluate the effectiveness and safety of the combination of Pembrolizumab (KEYTRUDA®) and the investigational drug, Metformin.

Patients will be randomized into one of two groups - either Arm A or Arm B. In Arm A, patients will receive pembrolizumab alone. In Arm B, patients will receive both pembrolizumab and metformin.

If patients are randomized to Arm A, they will be administered pembrolizumab (200 mg), by IV, every three weeks. After the first three doses, pembrolizumab dosing can be changed to 400mg IV every 6 weeks, at the treating physician's discretion. Pembrolizumab can be administered up to two years, if disease does not progress or have unacceptable toxicity. However, if the disease progresses the patient may continue on the study if they are clinically stable or clinically improved.

If patients are randomized to Arm B, they will be administered pembrolizumab (200 mg), by IV, every three weeks, plus metformin (500 mg), twice a day for nine weeks. Metformin will be taken in the morning and evening, 12hrs apart, with food. After the first three doses, pembrolizumab dosing can be changed to 400mg IV every 6 weeks, at the treating physician's discretion.

Discontinuation of treatment may be considered for patients who have attained a confirmed complete response that have been treated for at least 24 weeks with pembrolizumab and had at least two treatments with pembrolizumab beyond the date when the initial complete response was declared.

Patients will be followed for 5 years after removal from study or until death, whichever occurs first, through standard of care visits, phone call or by medical records review.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Have un-resectable (stage III) or advanced (stage IV) melanoma.
* Be 18 years of age or older on day of signing informed consent
* Have measurable disease based on RECIST 1.1. Patients without measurable disease may be included on study after discussion with the Sponsor, given that the primary endpoint of the study is Ki-67 of TIL (flow cytometry)
* Have biopsiable disease. Be willing to provide tissue from a newly obtained biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 30 days prior to initiation of treatment on Day 1.
* Patients may have received prior adjuvant therapy with anti-PD-1, anti-CTLA-4, or BRAF/MEK inhibitors.
* Patients may be immunotherapy treatment naïve in the advanced setting or may be on anti-PD-1 therapy with SD or PR for at least 12 weeks. Patients may have received ipilimumab plus nivolumab in the metastatic setting with SD or PR for at least 12 weeks on maintenance anti-PD1.
* Have a performance status of 0, 1 or 2 on the ECOG Performance Scale.
* Have a baseline HbA1c ≤ 6.4.
* Demonstrate adequate organ function. All screening labs should be performed within 14 days of treatment initiation.

  1. Absolute neutrophil count (ANC) ≥1,500 /mcL
  2. Platelets ≥100,000 / mcL
  3. Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  4. Serum creatinine OR Measured or calculateda creatinine clearance ≤1.5 X upper limit of normal (ULN) (GFR can also be used in place of creatinine or CrCl ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN)
  5. Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  6. AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  7. Albumin >2.5 mg/dL
  8. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants; Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Patients must be free of active brain metastases by contrast-enhanced CT/MRI scans within 2 weeks prior to starting the study drugs. If known to have prior brain metastases, must not have evidence of active (enlarging and/or symptomatic lesions) brain disease on MRI evaluation within 4 weeks from SRS or WBRT treatment.
* Patients who have received radiation may be enrolled if the treating physician determines that they have recovered from radiation and are not experiencing radiation related clinically significant adverse events.
* Female patients of child bearing potential must have a negative urine or serum pregnancy test within 7 days from the time of registration.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Has a current confirmed diagnosis of type 1 diabetes or type 2 diabetes that has been diagnosed by an HbA1c ≥6.5, or is on any hypoglycemic medications (insulin, metformin, etc). Patients with a screening HbA1c 6.5-7.0 may be included after discussion with the principal investigator. Patients currently on metformin will be excluded.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 (this excludes patients on anti-PD1) or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least two weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxineor physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic IV antibiotic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has a known history of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (hepatitis C virus [HCV] RNA [qualitative] is detected). Note: Without known history, testing only needs to be performed if there is clinical suspicion for Hepatitis B or C.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Ki-67 proliferation index in T cell | up to 4 years
  determine the cell cycle status

SECONDARY OUTCOMES:
Number of participants experiencing adverse events | up to 4 years
  Number of participants that received a combination of Pembrolizumab and Metformin who experience treatment-related adverse events as assessed by CTCAE v4.0
Hypoxia in the primary tumor by IHC Staining | up to 4 years
Mitochondrial functional restoration in Tumor Infiltrating Lymphocytes by mitochondrial mass | up to 4 years
  patients treated with metformin and pembrolizumab compared to pembrolizumab alone
Cell cycle status of peripheral blood T lymphocytes by Flow Cytometry | up to 4 years
  patients treated with pembrolizumab and metformin compared to patients treated with pembrolizumab alone
overall tumor response rate | up to 4 years
  patients treated with metformin and pembrolizumab compared to pembrolizumab alone, as measured by clinical tumor measurement and radiological tumor measurement on PET/CT scans.
Mitochondrial functional restoration in Tumor Infiltrating Lymphocytes by Seahorse metabolic profiling | up to 4 years
  patients treated with metformin and pembrolizumab compared to pembrolizumab alone

OTHER OUTCOMES:
Functional restoration of peripheral blood T lymphocytes | up to 4 years
Progression free survival | up to 5 years
Correlating hypoxia measurements in the tumor with FDG avidity on PET. | up to 4 years
MDSC in the tumor microenvironment and peripheral blood by flow cytometry. | up to 4 years
Melanoma tumor antigen specific T cell responses by flow cytometry. | up to 4 years
Overall survival | up to 5 years
Treg levels in the tumor microenvironment by flow cytometry | up to 4 years
Degree of mitochondrial functional restoration in TIL of patients treated with metformin and pembrolizumab compared to pembrolizumab alone | up to 4 years
  flow cytometry will be used to measure mitochondrial mass and glucose uptake in T cells

CONTACTS AND LOCATIONS:
Overall Officials: Yana Najjar, Md, Principal Investigator — Universtiy of Pittsburgh
Locations (1):
- Univ of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania, United States